CLINICAL TRIAL: NCT05871255
Title: Natural Topical Treatment for Vulvar and Vaginal Atrophy: a Single-center Prospective Observational Study
Brief Title: Natural Topical Treatment for Vulvar and Vaginal Atrophy
Status: Completed | Type: Observational
Sponsor: Dr. Amjad Khan (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor-Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Organization: Liaquat University of Medical & Health Sciences (Other)
Other Study IDs: 6407
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-05

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genitourinary syndrome of menopause (GSM) patients: Patients will apply the vaginal gel (ZG) for a total of 150 days of treatment. The application was daily for the first 12 days, then every 48 hours until the end of the study. Patients will be examined at baseline (T0), after 12 (T1), 57 (T2) and 150 (T3) days of treatment. Examination will include (1) Filling of a Female Sexual Distress Scale (FSDS) questionnaire and (2) Gynecology examination with colposcopy and pH test to evaluate vaginal elasticity, vaginal secretions, pH, mucosal epithelium, and vaginal hydration to calculate the Vaginal Health Index (VHI).
  Interventions: Other: Zantogin® Gel

INTERVENTIONS:
Other: Zantogin® Gel — Zantogin® Gel (ZG) is a multicomponent vaginal lubricant endowed with lenitive and anti-inflammatory properties, developed as class II medical device for the treatment of VVA.

SUMMARY:
Genitourinary syndrome of menopause (GSM) is a chronic and progressive syndrome characterized by a collection of genital and urinary signs and symptoms secondary to the state of hypoestrogenism related to menopause.

DETAILED DESCRIPTION:
The aim of this prospective observational study is to evaluate safety and efficacy of Zantogin® Gel (ZG) a class II medical device developed for intravaginal use in the treatment of signs and symptoms of post-menopausal vulvovaginal atrophy (VVA), in terms of improvement of objective parameters assessing vaginal health (Vaginal Health Index score) and subsequent patients' sexual quality of life (Female Sexual Distress Scale).

ELIGIBILITY:
Inclusion Criteria:

* Age between 45-65 years
* Menopause and symptomatic vulvovaginal atrophy (VVA) (vaginal dryness, dyspareunia, vaginal irritation, vaginal itching, dysuria)
* No previous treatment for VVA
* Informed written consent signed

Exclusion Criteria:

* Pregnancy
* Previous or concurrent neoplasms
* Uncompensated concomitant diseases (i.e., diabetes, cardiac diseases)
* Previous or concurrent Hormone replacement therapy (HRT) or radiotherapy or chemotherapy.

Ages: 45 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is related to a health condition only occurs in females
Study Population: Same as the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in vaginal health index score | 5.5 months
  Scale score range is 5-25. The minimum 5 points core indicates severe vulvovaginal atrophy and the maximum total score of 25 points indicates no clinical signs of vulvovaginal atrophy.
Change in Female Sexual Distress Scale (FSD) | 5.5 months
  A score of ≥11 effectively discriminates between women with FSD and no FSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Maternal-Fetal Medicine at Policlinico Umberto, Rome, Italy